CLINICAL TRIAL: NCT01350310
Title: Intramyocardial Stem Cell Therapy in Patients With Dilated Cardiomyopathy
Brief Title: Safety and Efficacy Study of Intramyocardial Stem Cell Therapy in Patients With Dilated Cardiomyopathy
Acronym: NOGA-DCM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Collaborators: The Methodist Hospital Research Institute (Other); Stanford University (Other)
Responsible Party: Principal Investigator, Bojan Vrtovec, Prof. Dr. Bojan Vrtovec, dr. med., University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NOGA-DCM
Record Dates: First submitted 2011-05-06; First posted 2011-05-09 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Dilated Cardiomyopathy; Chronic Heart Failure
Keywords: Heart failure; Dilated cardiomyopathy; Stem cells
MeSH Terms: conditions — Cardiomyopathy, Dilated; Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Intramyocardial Injections (Experimental): Peripheral blood stem cells will be mobilised by daily subcutaneous injections of filgrastim; CD34+ cells will be collected via apheresis and labelled with technetium. Electromechanical mapping will be used to identify viable myocardium and intramyocardial injections in the target areas will be performed with NOGA catheter. Nuclear imaging for quantitation of myocardial retention rates of labeled cells will be performed at 2 and 18 hours after the procedure.
  Interventions: Procedure: Intramyocardial injection
- Intracoronary Injections (Active Comparator): Peripheral blood stem cells will be mobilised by daily subcutaneous injections of filgrastim; CD34+ cells will be collected via apheresis and labelled with technetium. Patients will undergo myocardial perfusion scintigraphy and CD34+ cells will be injected intracoronary in the artery supplying segments of reduced viability. Nuclear imaging for quantitation of myocardial retention rates of labeled cells will be performed at 2 and 18 hours after the procedure.
  Interventions: Procedure: Intracoronary injection
- Ischemic heart disease (Active Comparator): Peripheral blood stem cells will be mobilised by daily subcutaneous injections of filgrastim; CD34+ cells will be collected via apheresis and labelled with technetium. Electromechanical mapping will be used to identify viable myocardium and intramyocardial injections in the target areas will be performed with NOGA catheter. Nuclear imaging for quantitation of myocardial retention rates of labeled cells will be performed at 2 and 18 hours after the procedure
  Interventions: Procedure: Intramyocardial injection

INTERVENTIONS:
Procedure: Intramyocardial injection — Electromechanical mapping will be used to identify viable myocardium (unipolar voltage >6.9 mV) and intramyocardial injections in the target areas will be performed with NOGA catheter (25 injections of 0.3 cc).
  Arms: Intramyocardial Injections
Procedure: Intracoronary injection — Patients will undergo myocardial perfusion scintigraphy for myocardial viability assessment. Microcatheter will be placed in the mid segment of the coronary artery supplying the segments of reduced tracer accumulation and repeated intracoronary injections of stem cell solution will be performed.
  Arms: Intracoronary Injections
Procedure: Intramyocardial injection — Procedure/Surgery: Intramyocardial injection Electromechanical mapping will be used to identify viable myocardium (unipolar voltage >6.9 mV) and intramyocardial injections in the target areas will be performed with NOGA catheter (25 injections of 0.3 cc).
  Arms: Ischemic heart disease

SUMMARY:
BACKGROUND. In patients with non-ischemic dilated cardiomyopathy, intracoronary stem cell transplantation has been shown to improve exercise capacity, reduce ventricular remodelling and improve 1-year survival. Pre-clinical data demonstrate that stem cell effects on the diseased heart can be further enhanced by direct intramyocardial delivery route.

AIMS.

1. To evaluate safety and efficacy of intramyocardial stem cell therapy in patients with non-ischemic dilated cardiomyopathy.
2. To directly compare clinical effects of intracoronary and intramyocardial stem cell delivery.

METHODS. Of 60 patients with dilated cardiomyopathy, 30 will be randomized to intramyocardial transplantation of CD34+ cells (Study Group), and 30 will receive intracoronary stem cell therapy (Control Group). In both groups peripheral blood stem cells will be mobilised by daily subcutaneous injections of filgrastim; CD34+ cells will be collected via apheresis and labelled with technetium. In the Study Group electromechanical mapping will be used to identify viable myocardium and intramyocardial injections in the target areas will be performed with NOGA catheter. In the Control group patients will undergo myocardial perfusion scintigraphy and CD34+ cells will be injected intracoronary in the artery supplying segments of reduced viability. Patients will be followed for 1 year. Primary endpoints will include changes in left ventricular ejection fraction and left ventricular dimensions (measured by echocardiography). Secondary endpoints will include changes in exercise capacity and changes in NT-proBNP values.

HYPOTHESES.

1. At 1 year, intramyocardial stem cell therapy will be associated with improved left ventricular ejection fraction, reduced left ventricular dimensions, improved exercise capacity and reduced levels of NT-proBNP.
2. Beneficial effects of intramyocardial stem cell therapy will be superior to those observed with intracoronary stem cell delivery.

ELIGIBILITY:
Inclusion Criteria:

* Established dg. of dilated CMP (defined according to ESC position statement - absence of any stenotic lesions on coronary angiography, no congenital heart disease, no primary valve disease on echocardiography, and no history of hypertension or alcohol abuse1)
* left ventricular ejection fraction < 30%
* NYHA functional class III or IV for at least 3 months before referral
* Optimal medical management for at least 6 months

Exclusion Criteria:

* Left ventricular aneurysm or thrombus
* Hematologic disease
* Multiorgan failure
* Active malignancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2011-03; Primary Completion 2014-08 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Changes in left ventricular ejection fraction and dimensions | 1 year
  Standard 2D and Doppler echocardiography will be performed at baseline, and repeated at 1 month, 3 months, 6 months and 1 year after the procedure. Left ventricular ejection fraction will be measured using Simpson's method and left ventricular end-systolic and end-diastolic dimensions will be measured according to standard echocardiography protocol.

SECONDARY OUTCOMES:
Changes in exercise capacity | 1 year
  Exercise capacity will be evaluated with 6-minute walk test at baseline, and again at 1,3,6 and 12 months after the procedure.
Change in NT-proBNP levels | 1 year
  Plasma levels of NT-proBNP will be measured at baseline, and again at 1, 3, 6 and 12 months after the procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- UMC Ljubljana, Ljubljana, Slovenia

REFERENCES:
- [Derived] Lezaic L, Socan A, Poglajen G, Peitl PK, Sever M, Cukjati M, Cernelc P, Wu JC, Haddad F, Vrtovec B. Intracoronary transplantation of CD34(+) cells is associated with improved myocardial perfusion in patients with nonischemic dilated cardiomyopathy. J Card Fail. 2015 Feb;21(2):145-52. doi: 10.1016/j.cardfail.2014.11.005. Epub 2014 Nov 18. PMID 25459687
- [Derived] Poglajen G, Sever M, Cukjati M, Cernelc P, Knezevic I, Zemljic G, Haddad F, Wu JC, Vrtovec B. Effects of transendocardial CD34+ cell transplantation in patients with ischemic cardiomyopathy. Circ Cardiovasc Interv. 2014 Aug;7(4):552-9. doi: 10.1161/CIRCINTERVENTIONS.114.001436. Epub 2014 Aug 5. PMID 25097199
- [Derived] Vrtovec B, Poglajen G, Lezaic L, Sever M, Socan A, Domanovic D, Cernelc P, Torre-Amione G, Haddad F, Wu JC. Comparison of transendocardial and intracoronary CD34+ cell transplantation in patients with nonischemic dilated cardiomyopathy. Circulation. 2013 Sep 10;128(11 Suppl 1):S42-9. doi: 10.1161/CIRCULATIONAHA.112.000230. PMID 24030420
- [Derived] Vrtovec B, Poglajen G, Lezaic L, Sever M, Domanovic D, Cernelc P, Socan A, Schrepfer S, Torre-Amione G, Haddad F, Wu JC. Effects of intracoronary CD34+ stem cell transplantation in nonischemic dilated cardiomyopathy patients: 5-year follow-up. Circ Res. 2013 Jan 4;112(1):165-73. doi: 10.1161/CIRCRESAHA.112.276519. Epub 2012 Oct 12. PMID 23065358